CLINICAL TRIAL: NCT00407537
Title: A Cluster Randomized Trial On Cardiovascular Risk Factor Management: Caduet Versus Usual Care In Subjects With Hypertension And Additional Cardiovascular Risk Factors In Clinical Practice
Brief Title: Caduet vs Usual Care in Subjects With Hypertension and Additional Risk Factors
Acronym: CRUCIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3841047
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hypercholesterolemia
MeSH Terms: conditions — Hypertension; Hypercholesterolemia | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caduet (Experimental): Open label caduet added to usual care regimen followed by investigators.
  Interventions: Drug: Amlodipine besylate/atorvastatin calcium single pill combination

INTERVENTIONS:
Drug: Amlodipine besylate/atorvastatin calcium single pill combination — Open label amlodipine besylate/atorvastatin calcium single pill combination at multiple doses: 5/10, 10/10, 5/20, 10/20 mg prescribed at the investigator's discretion

SUMMARY:
To investigate whether a Caduet based treatment strategy might result in greater reduction in total cardiovascular risk as compared to usual care in subjects with hypertension and additional risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension with three additional risks factors (for example: smoking, type 2 diabetes, family history of early heart disease, history of stroke, age over 55 (men) and 65 (women)

Exclusion Criteria:

* Subjects currently receiving a statin or stopped statin within 6 months prior to enrollment.
* Subjects with a history of myocardial infarction and subjects with coronary bypass graft or intra-coronary interventions.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1531 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- Costa Rica (3):
  - Pfizer Investigational Site, Desamparados, Provincia de San José
  - Pfizer Investigational Site, Heredia
  - Pfizer Investigational Site, San José
- Croatia (10):
  - Pfizer Investigational Site, Breznički Hum
  - Pfizer Investigational Site, Crikvenica
  - Pfizer Investigational Site, Čakovec
  - Pfizer Investigational Site, Karlovac
  - Pfizer Investigational Site, Rijeka
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Sveti Križ Začretje
  - Pfizer Investigational Site, Špišić-Bukovica
  - Pfizer Investigational Site, Varaždin
  - Pfizer Investigational Site, Zagreb
- Czechia (11):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Klatovy
  - Pfizer Investigational Site, Kralupy nad Vltavou
  - Pfizer Investigational Site, Lanškroun
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Pelhřimov
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Průhonice
  - Pfizer Investigational Site, Ústí nad Labem
  - Pfizer Investigational Site, Vratimov
  - Pfizer Investigational Site, Zlín
- Dominican Republic (2):
  - Pfizer Investigational Site, San Cristóbal
  - Pfizer Investigational Site, Santo Domingo
- Indonesia (7):
  - Pfizer Investigational Site, Cilandak, Jakarta Selatan
  - Pfizer Investigational Site, Bandung
  - Pfizer Investigational Site, Jakarta
  - Pfizer Investigational Site, Semarang
  - Pfizer Investigational Site, Surabaya
  - Pfizer Investigational Site, Tangerang
  - Pfizer Investigational Site, Tanggerang
- Jordan (2):
  - Pfizer Investigational Site, Amman
  - Pfizer Investigational Site, Irbid
- Kuwait (2):
  - Pfizer Investigational Site, Kuwait City
  - Pfizer Investigational Site, Sasat
- Lebanon (2):
  - Pfizer Investigational Site, Beirut
  - Pfizer Investigational Site, Byblos
- Malaysia (6):
  - Pfizer Investigational Site, Kuala Pilah, Negeri Sembilan
  - Pfizer Investigational Site, Seremban, Negeri Sembilan
  - Pfizer Investigational Site, Batu Caves, Selangor
  - Pfizer Investigational Site, Petaling Jaya, Selangor
  - Pfizer Investigational Site, Butterworth
  - Pfizer Investigational Site, Kuala Lumpur
- Mexico (5):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Toluca, State of Mexico
  - Pfizer Investigational Site, Durango
  - Pfizer Investigational Site, San Luis Potosí City
- Pfizer Investigational Site, Panama City, Panama
- Philippines (5):
  - Pfizer Investigational Site, San Juan City, National Capital Region
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Marikina City
  - Pfizer Investigational Site, Quezon City
- Russia (5):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
  - Pfizer Investigational Site, Volgograd
  - Pfizer Investigational Site, Voronezh
- Pfizer Investigational Site, Riyadh, Saudi Arabia
- South Korea (9):
  - Pfizer Investigational Site, Wŏnju, Gangwon-do
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Suwon
- Taiwan (4):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, Rajthevee, Bangkok
  - Pfizer Investigational Site, Saimai, Bangkok
  - Pfizer Investigational Site, Bangkok
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
- United Arab Emirates (3):
  - Pfizer Investigational Site, Abu Dhabi
  - Pfizer Investigational Site, Al Ain City
  - Pfizer Investigational Site, Dubai
- Venezuela (3):
  - Pfizer Investigational Site, Naguanagua/Valencia, Carabobo
  - Pfizer Investigational Site, Valencia, Carabobo
  - Pfizer Investigational Site, Caracas, Dtto Capital/Municipio Libertador

REFERENCES:
- [Derived] Cho EJ, Kim JH, Sutradhar S, Yunis C, Westergaard M; CRUCIAL Trial Investigators. Proactive multifactorial intervention strategy reduces the risk of cardiovascular disease estimated with region-specific risk assessment models in Pacific Asian patients participating in the CRUCIAL trial. J Korean Med Sci. 2013 Dec;28(12):1741-8. doi: 10.3346/jkms.2013.28.12.1741. Epub 2013 Nov 26. PMID 24339703
- [Derived] Hradec J, Zamorano J, Sutradhar S. Post hoc analysis of the Cluster Randomized Usual Care versus Caduet Investigation Assessing Long-term risk (CRUCIAL) trial. Curr Med Res Opin. 2013 Jun;29(6):589-96. doi: 10.1185/03007995.2013.783795. Epub 2013 Apr 3. PMID 23464930
- [Derived] Kim JH, Zamorano J, Erdine S, Pavia A, Al-Khadra A, Sutradhar S, Yunis C; CR UCIAL Investigators. Proactive cardiovascular risk management versus usual care in patients with and without diabetes mellitus: CRUCIAL trial subanalysis. Postgrad Med. 2012 Jul;124(4):41-53. doi: 10.3810/pgm.2012.07.2565. PMID 22913893
- [Derived] Zamorano J, Erdine S, Pavia A, Kim JH, Al-Khadra A, Westergaard M, Sutradhar S, Yunis C; CRUCIAL Investigators. Proactive multiple cardiovascular risk factor management compared with usual care in patients with hypertension and additional risk factors: the CRUCIAL trial. Curr Med Res Opin. 2011 Apr;27(4):821-33. doi: 10.1185/03007995.2011.555754. Epub 2011 Feb 10. PMID 21306285
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841047&StudyName=Caduet%20vs%20Usual%20Care%20in%20Subjects%20with%20Hypertension%20and%20Additional%20Risk%20Factors

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cluster randomized study: the unit of randomization was the investigator, ie, participants were screened before the investigator was randomized. A total of 136 sites were cluster randomized.
Pre-assignment Details: Prior to group assignment of investigators (who were the unit of randomization), participants were consented and screened for enrollment eligibility; participant selection for enrollment took place before investigator assignment. A total of 1,531 participants were enrolled and attended baseline visit; 1,461 participants received treatment.
Groups:
- Caduet: Open label amlodipine besylate/atorvastatin calcium (Caduet) single pill combination at multiple doses: 5/10, 10/10, 5/20, 10/20 mg prescribed at the investigator's discretion.
- Usual Care: Full choice of any locally approved (and not contra indicated) anti-hypertensive and/or lipid lowering drugs, including, but not limited to amlodipine and atorvastatin, according to local clinical practice.
Period: Overall Study
Arm/Group | Caduet | Usual Care
Started | 779 | 682 (4 participants assigned to Caduet treatment received usual care only during the study)
Eligible for Efficacy Analysis | 760 | 657
Completed | 686 | 638
Not Completed | 93 | 44
Not completed — Death | 5 | 2
Not completed — Adverse Event | 36 | 0
Not completed — Lost to Follow-up | 12 | 19
Not completed — Other | 6 | 7
Not completed — Withdrawal by Subject | 34 | 16

BASELINE CHARACTERISTICS:
Groups:
- Caduet as Assigned: Open label amlodipine besylate/atorvastatin calcium (Caduet) single pill combination at multiple doses: 5/10, 10/10, 5/20, 10/20 mg prescribed at the investigator's discretion.
- Usual Care as Assigned: Full choice of any locally approved (and not contra indicated) anti-hypertensive and/or lipid lowering drugs, including, but not limited to amlodipine and atorvastatin, according to local clinical practice.
- Total: Total of all reporting groups
Arm/Group | Caduet as Assigned | Usual Care as Assigned | Total
Number analyzed (Participants) | 783 | 678 | 1461
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0
  18 to 44 years | 58 | 55 | 113
  45 to 64 years | 450 | 361 | 811
  > = 65 years | 275 | 262 | 537
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 368 | 334 | 702
  Male | 415 | 344 | 759

OUTCOME MEASURES:

1. Primary Outcome: Framingham 10-year Risk of Total Coronary Heart Disease (CHD) at Month 12
Description: Framingham prediction of 10-year risk of CHD: Gender-specific prediction equations formulated to predict CHD risk according to age, diabetes, smoking, blood pressure categories, and total cholesterol and low density lipoprotein (LDL) cholesterol categories. The coefficients were used to derive the score calculated at the end of study treatment (Month 12).
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) included all subjects, in either treatment group, who had blood pressure and lipid data from at least 1 follow-up visit. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 748 | 655
percent risk | 12.5 (8.26) | 16.3 (10.51)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; It was estimated that each study site would on average complete 8 evaluable participants, therefore enrolling 164 sites, 1968 participants would provide at least 90% power to detect a 10% relative reduction in the 10-year predicted risk of total CHD at 12 months (as calculated from the Framingham model) from the control arm based on a two-sided t-test with a 5% significance level; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — Value at a given visit as response. Baseline value, country, and treatment were used as fixed effect and site was used as a random effect and a compound-symmetry (CS) variance-covariance matrix was used for subjects from the same site; LSMean difference = -4.72, 95% CI 2-sided [-5.55 to -3.89] — Value at a given visit as response. Baseline value, country, and treatment were used as fixed effect and site was used as a random effect and a compound-symmetry (CS) variance-covariance matrix was used for subjects from the same site

2. Secondary Outcome: Framingham 10-year Risk of Total CHD at Month 4
Description: Framingham prediction of 10-year risk of CHD: Gender-specific prediction equations formulated to predict CHD risk according to age, diabetes, smoking, blood pressure categories, and total cholesterol and low density lipoprotein (LDL) cholesterol categories. The coefficients were used to derive the score calculated after 4 months of treatment (Month 4).
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 745 | 637
percent risk | 12.5 (7.96) | 16.3 (10.80)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -4.76, 95% CI 2-sided [-5.58 to -3.93] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: European Systematic COronary Risk Evaluation (SCORE) 10-year Risk of Fatal Cardiovascular Disease (CVD) at Month 12
Description: European SCORE: designed to measure cardiovascular disease mortality; computed using age, gender, whether a person lives in a low risk or high risk region, measured total cholesterol, measured HDL cholesterol, systolic blood pressure, and current smoking status. The coefficients were used to derive the score calculated after 12 months of study treatment (Month 12).
Time Frame: Baseline, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 748 | 655
percent risk | 3.0 (2.89) | 3.7 (3.69)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.97, 95% CI 2-sided [-1.23 to -0.72] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: European SCORE 10-year Risk of Fatal CVD at Month 4
Description: European SCORE: designed to measure cardiovascular disease mortality; computed using age, gender, whether a person lives in a low risk or high risk region, measured total cholesterol, measured HDL cholesterol, systolic blood pressure, and current smoking status. The coefficients were used to derive the score calculated after 4 months of study treatment (Month 4).
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 745 | 637
percent risk | 3.1 (3.13) | 3.7 (3.69)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -0.88, 95% CI 2-sided [-1.16 to -0.59] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Framingham 10-year Risk of Stroke at Month 12
Description: Stroke risk calculated from the Framingham risk for CVD (CHD, stroke, intermittent claudication, congestive heart failure) multiplied by a gender-specific "calibration factor" for the stroke component risk. Coefficients were used to derive the score calculated at the end of study treatment (Month 12).
Time Frame: Baseline, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 748 | 655
percent risk | 3.7 (2.25) | 4.9 (2.87)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.35, 95% CI 2-sided [-1.56 to -1.15] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Framingham 10-year Risk of Stroke at Month 4
Description: as for outcome 5
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 745 | 637
percent risk | 3.7 (2.21) | 4.9 (2.81)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 1, analysis 1]; LSMean difference = -1.35, 95% CI 2-sided [-1.57 to -1.14] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Framingham 10-year Risk of Developing Total CHD
Description: Framingham prediction of 10-year risk of CHD: Gender-specific prediction equations formulated to predict CHD risk according to age, diabetes, smoking, blood pressure categories, and total cholesterol and low density lipoprotein (LDL) cholesterol categories. Change from baseline calculated as mean at observation minus mean at Baseline.
Time Frame: Baseline, Month 4, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
percent risk
  Month 4 | -7.2705 [-7.90 to -6.64] | -2.5155 [-3.19 to -1.84]
  Month 12 | -7.2374 [-7.87 to -6.61] | -2.5167 [-3.19 to -1.84]

8. Secondary Outcome: Change From Baseline European SCORE 10-year Risk of Developing Fatal CVD
Description: European SCORE: designed to measure cardiovascular disease mortality; computed using age, gender, whether a person lives in a low risk or high risk region, measured total cholesterol, measured HDL cholesterol, systolic blood pressure, and current smoking status. Change from baseline calculated as mean at observation minus mean at Baseline.
Time Frame: Baseline, Month 4, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent risk
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 748 | 655
percent risk
  Month 4 | -1.8438 [-2.06 to -1.63] | -0.9678 [-1.20 to -0.74]
  Month 12 | -1.9693 [-2.16 to -1.77] | -0.9963 [-1.21 to -0.79]

9. Secondary Outcome: Mean Systolic and Diastolic Blood Pressure at Month 4
Time Frame: Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 759 | 657
mmHg
  Systolic | 133.5 (14.32) | 134.5 (14.96)
  Diastolic | 80.7 (8.74) | 81.1 (9.32)

10. Secondary Outcome: Mean Systolic and Diastolic Blood Pressure at Month 12
Time Frame: Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mmHg
  Systolic | 130.6 (13.84) | 134.3 (15.21)
  Diastolic | 79.2 (8.39) | 81.1 (9.27)

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Month 4
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 759 | 657
mmHG | -15.3088 [-17.02 to -13.60] | -12.1619 [-14.00 to -10.32]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.007, Mixed-effect linear model; Mean Difference (Final Values) = -3.15, 95% CI 2-sided [-5.42 to -0.88]

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Month 4
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHG
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 759 | 657
mmHG | -8.3024 [-9.24 to -7.36] | -6.6908 [-7.70 to -5.68]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.011, Mixed-effect linear model; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-2.86 to -0.37]

13. Secondary Outcome: Change From Baseline in SBP at Month 12
Time Frame: Baseline, Month 12
Population: FAS, number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mmHg | -18.2409 [-19.94 to -16.55] | -12.4903 [-14.32 to -10.66]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model; Mean Difference (Final Values) = -5.75, 95% CI 2-sided [-8.00 to -3.50]

14. Secondary Outcome: Change From Baseline in DBP at Month 12
Time Frame: Baseline, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing to data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mmHg | -10.0128 [-10.96 to -9.07] | -6.8429 [-7.86 to -5.83]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model; Mean Difference (Final Values) = -3.17, 95% CI 2-sided [-4.42 to -1.92]

15. Secondary Outcome: Mean Lipid Parameters at Month 4
Description: Mean Total Cholesterol (TC), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), and Triglyceride blood concentrations.
Time Frame: Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mg/dL
  TC | 156.0 (34.14) | 195.2 (37.03)
  LDL | 80.9 (28.47) | 116.4 (32.47)
  HDL | 47.6 (13.93) | 46.8 (13.49)
  Triglycerides | 143.5 (83.26) | 164.8 (95.74)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; TC; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — Baseline value, country, and treatment were used as fixed effect and site was used as a random effect and a compound-symmetry (CS) variance-covariance matrix was used for subjects from the same site; Mean Difference (Final Values) = -38.94, 95% CI 2-sided [-43.71 to -34.17]
Statistical Analysis 2: Comparison: Caduet vs Usual Care; LDL; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -35.31, 95% CI 2-sided [-39.64 to -30.99]
Statistical Analysis 3: Comparison: Caduet vs Usual Care; HDL; Test type: Superiority or Other; p = 0.087, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [-0.14 to 2.13]
Statistical Analysis 4: Comparison: Caduet vs Usual Care; Triglycerides; Test type: Superiority or Other; p < 0.001, Mixed-effects linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -23.65, 95% CI 2-sided [-32.60 to -14.70]

16. Secondary Outcome: Mean Lipid Parameters at Month 12
Description: as for outcome 15
Time Frame: Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mg/dL
  TC | 163.3 (38.42) | 196.6 (36.36)
  LDL | 87.1 (32.40) | 117.3 (31.57)
  HDL | 47.3 (13.48) | 47.1 (13.61)
  Triglycerides | 151.5 (98.61) | 166.4 (98.53)
Statistical Analysis 1: Comparison: Caduet vs Usual Care; TC; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -33.07, 95% CI 2-sided [-37.57 to -28.56]
Statistical Analysis 2: Comparison: Caduet vs Usual Care; LDL; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -29.83, 95% CI 2-sided [-33.70 to -25.95]
Statistical Analysis 3: Comparison: Caduet vs Usual Care; HDL; Test type: Superiority or Other; p = 0.379, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.71 to 1.86]
Statistical Analysis 4: Comparison: Caduet vs Usual Care; Triglycerides; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -18.27, 95% CI 2-sided [-28.72 to -7.81]

17. Secondary Outcome: Change From Baseline in Lipid Parameters at Month 4
Description: Mean Total Cholesterol (TC), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), and Triglyceride blood concentrations. Change from baseline measured as mean at Month 4 minus mean at Baseline.
Time Frame: Baseline, Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 752 | 630
mg/dL
  TC | -42.7542 [-46.35 to -39.15] | -3.8144 [-7.75 to 0.12]
  LDL | -38.2765 [-41.52 to -35.03] | -2.9628 [-6.50 to 0.58]
  HDL | -0.2060 [-1.07 to 0.65] | -1.1978 [-2.13 to -0.26]
  Triglycerides | -20.5645 [-27.30 to -13.83] | 3.0828 [-4.26 to 10.43]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; TC; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -38.94, 95% CI 2-sided [-43.71 to -34.17]
Statistical Analysis 2: Comparison: Caduet vs Usual Care; LDL; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -35.31, 95% CI 2-sided [-39.64 to -30.99]
Statistical Analysis 3: Comparison: Caduet vs Usual Care; HDL; Test type: Superiority or Other; p = 0.087, mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [-0.14 to 2.13]
Statistical Analysis 4: Comparison: Caduet vs Usual Care; Triglycerides; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -23.65, 95% CI 2-sided [-32.60 to -14.70]

18. Secondary Outcome: Change From Baseline in Lipid Parameters at Month 12
Description: as for outcome 15
Time Frame: Baseline, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
mg/dL
  TC | -37.1024 [-40.52 to -33.69] | -4.0368 [-7.71 to -0.36]
  LDL | -33.2420 [-36.17 to -30.32] | -3.4168 [-6.58 to -0.25]
  HDL | -0.4339 [-1.41 to 0.54] | -1.0105 [-2.06 to 0.04]
  Triglycerides | -15.2270 [-23.12 to -7.33] | 3.0398 [-5.51 to 11.59]
Statistical Analysis 1: Comparison: Caduet vs Usual Care; Total cholesterol; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -33.07, 95% CI 2-sided [-37.57 to -28.56]
Statistical Analysis 2: Comparison: Caduet vs Usual Care; LDL; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -29.83, 95% CI 2-sided [-33.70 to -25.95]
Statistical Analysis 3: Comparison: Caduet vs Usual Care; HDL; Test type: Superiority or Other; p = 0.379, mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.71 to 1.86]
Statistical Analysis 4: Comparison: Caduet vs Usual Care; Triglycerides; Test type: Superiority or Other; p < 0.001, Mixed-effect linear model — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = -18.27, 95% CI 2-sided [-28.72 to -7.81]

19. Secondary Outcome: Percentage of Participants at Conventional Treatment Goals According to Global and Local Guidelines for Blood Pressure at 4 and 12 Months
Description: Goals set at <140/90 mmHg according to the seventh Joint National Committee (JNC) on prevention, detection, evaluation, and treatment of high blood pressure and <140/90 mm Hg or <130/80 mm Hg for diabetics ccording to the European Society of Cardiology (ESC) guidelines.
Time Frame: Month 4, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Number; unit: percentage of participants
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
percentage of participants
  JNC Month 4 | 65.2 | 62.6
  JNC Month 12 | 76.1 | 60.6
  ESC Month 4 | 48.6 | 46.0
  ESC Month 12 | 58.2 | 47.5

20. Secondary Outcome: Percentage of Participants at Conventional Treatment Goals According to Global and Local Guidelines for LDL at 4 and 12 Months
Description: Goal set at <100 mg/dL according to the United States (US) National Cholesterol Education Program Adult Treatment Panel 3 and at <80 mg/dL according to the European (EU) Society of Cardiology guidelines.
Time Frame: Month 4, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
Percentage of participants
  US Month 4 | 77.3 | 28.2
  US Month 12 | 71.9 | 28.8
  EU Month 4 | 52.4 | 13.3
  EU Month 12 | 46.7 | 11.5

21. Secondary Outcome: Number of Participants With Lipid and Antihypertensive Treatments Used at 4 and 12 Months
Description: Treatments indicative of prescribed medications other than study provided Caduet.
Time Frame: Month 4, Month 12
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Number; unit: participants
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
participants
  Month 4: anti-hypertensive and/or lipid lowering | 648 | 642
  Month 4: anti-hypertensive | 647 | 637
  Month 4: lipid lowering | 45 | 202
  Month 4: anti-hypertensive and lipid lowering | 44 | 197
  Month 12: anti-hypertensive and/or lipid lowering | 655 | 642
  Month 12: anti-hypertensive | 654 | 638
  Month 12: lipid lowering | 46 | 208
  Month 12: anti-hypertensive and lipid lowering | 45 | 204

22. Secondary Outcome: Number of Participants With Increase of Treatment Dosages After 4 Months.
Description: Treatments indicative of prescribed medications other than study provided Caduet.
Time Frame: Month 4
Population: FAS. Number of participants analyzed refers to number of participants contributing data.
Measure: Number; unit: Participants
Arm/Group | Caduet | Usual Care
Number analyzed (Participants) | 760 | 657
Participants
  Increased dose | 30 | 90
  increased dose of anti-hypertensive medications | 30 | 88
  increased dose of lipid lowering medications | 0 | 2
  increase in either medication | 4 | 45
  increase in both medications | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Caduet | Usual Care
Serious Adverse Events (participants affected / at risk) | 51/779 | 22/682
Other Adverse Events (participants affected / at risk) | 356/779 | 289/682
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caduet (N=779) | Usual Care (N=682)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Normal tension glaucoma (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Upper motor neurone lesion (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Choluria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caduet (N=779) | Usual Care (N=682)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 9 | 5
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 5 | 3
Chalazion (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 4 | 3
Conjunctivitis allergic (Eye disorders) | 0 | 2
Diabetic retinopathy (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Posterior capsule opacification (Eye disorders) | 2 | 0
Refraction disorder (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 3 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7
Colitis (Gastrointestinal disorders) | 0 | 2
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 9 | 4
Diabetic enteropathy (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 10
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 6
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gingival erythema (Gastrointestinal disorders) | 1 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 3
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 3
Periodontitis (Gastrointestinal disorders) | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 3 | 1
Chest discomfort (General disorders) | 4 | 4
Chest pain (General disorders) | 16 | 10
Drug ineffective (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 3
Generalised oedema (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Oedema (General disorders) | 11 | 1
Oedema peripheral (General disorders) | 52 | 11
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Swelling (General disorders) | 0 | 1
Tenderness (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 3
Hepatic steatosis (Hepatobiliary disorders) | 1 | 3
Allergy to arthropod sting (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 5
Bacterial infection (Infections and infestations) | 2 | 0
Borrelia infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 12 | 15
Bronchitis viral (Infections and infestations) | 0 | 1
Campylobacter intestinal infection (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 4 | 2
Eczema infected (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 3
Gingival infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 7 | 3
Labyrinthitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 22 | 10
Onychomycosis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 6 | 13
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 7
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 14
Urethritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 6
Urogenital infection fungal (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 2 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 3 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 2
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 2
Blood creatine increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 15 | 5
Blood creatinine increased (Investigations) | 6 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 8 | 3
Blood potassium decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 3
Blood pressure abnormal (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 2
Blood triglycerides increased (Investigations) | 11 | 14
Blood urea increased (Investigations) | 2 | 1
Blood uric acid increased (Investigations) | 0 | 2
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
High density lipoprotein increased (Investigations) | 1 | 0
Lipids increased (Investigations) | 0 | 1
Platelet aggregation increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 11
Food intolerance (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 12
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 4
Hypo HDL cholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 6
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 8
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Senile osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Balance disorder (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 17 | 9
Dizziness postural (Nervous system disorders) | 0 | 2
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 23 | 15
Hypoaesthesia (Nervous system disorders) | 8 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Nerve root lesion (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 3 | 1
Tension headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 5
Bruxism (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 8 | 11
Neurosis (Psychiatric disorders) | 0 | 1
Tic (Psychiatric disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Circumcision (Surgical and medical procedures) | 1 | 0
Intraocular lens implant (Surgical and medical procedures) | 1 | 1
Lipoma excision (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 6 | 12
Hypotension (Vascular disorders) | 9 | 4
Intermittent claudication (Vascular disorders) | 2 | 0
Labile blood pressure (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Venous insufficiency (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.